CLINICAL TRIAL: NCT02015702
Title: Interventions to Increase Physician Effectiveness and Acceptance of a Electronic Health Record System
Brief Title: Educational Intervention to Increase Physician Satisfaction and Effectiveness With a New Electronic Health Record
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Reading Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ReadingHMC-IRB-045-12
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2013-12

CONDITIONS: Attitude of Health Personnel
Keywords: Physicians; Electronic Health Record; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-on-one physician training (Experimental): One-on-one physician training Physicians in the experimental arm were visited by a instructing physician at a computer while performing clinical duties who had observed others to identify best practices. Instructors watched subjects' work, looking for a specific tip that could be applied to the current work, then demonstrated the tip, and answered any questions the subject had about using or applying this new technique .
  Interventions: Other: One-on-one physician training; Other: Usual training
- Usual training (Active Comparator): Usual training. This group will get the usual specified training for learning to use our electronic health record. Both groups received 12 hours of EPIC classroom training, exposure to the EPIC e-learning modules, user acceptability testing classes, and unlimited time on the EPIC 'playground', a site to practice on virtual patients. All had 90 days of elbow support with an EPIC-training non-physician technician, who were visible and available on all inpatient wards, as well as access to a physician-only support line available at all hours.
  Interventions: Other: Usual training

INTERVENTIONS:
Other: One-on-one physician training — Physicians in the experimental arm were visited by a instructing physician at a computer while performing clinical duties who had observed others to identify best practices. Instructors watched subjects' work, looking for a specific tip that could be applied to the current work, then demonstrated the tip, and answered any questions the subject had about using or applying this new technique .
  Arms: One-on-one physician training
Other: Usual training — Usual training included online e-modules, 12 hours of classroom time, practice in the EPIC Playground, user acceptability training classes,non-physician technical support on all of the floors, and a physician-only help line.

SUMMARY:
This study was intended to test the effects of adding a one-on-one educational intervention taught by a physician to a physician during their clinical work to improve their acceptance and satisfaction with a new inpatient electronic health record and ordering system.

DETAILED DESCRIPTION:
This study was a randomized, parallel , non- blinded controlled trial of real-time, focused educational interventions in an intervention arm compared with usual training and support in the control arm. Improvement in performance, defined as the time between opening and closing a progress note, and number of notes completed after shift , were the primary outcomes. Physician satisfaction was a secondary outcome. Participants from one 550-bed Academic Independent Medical Center were invited to participate if they were full-time hospitalists or residents in internal medicine with no prior experience with the EPIC electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* Internal Medicine physicians and resident physicians with inpatient clinical duties at the time of the EPIC electronic health record go-live (Feb 4, 2013)

Exclusion Criteria:

* Physicians whose duties did not include regular admissions and discharge of patients
* Physicians whose work was limited to teaching
* Physicians with prior experience in using EPIC systems for inpatient care .
* Physician assistants and nurse practitioners

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2014-01-14 (Actual)

PRIMARY OUTCOMES:
Time to complete a progress note | within 1 week of note completion
  the primary outcome measure will be time to complete a progress note. this is defined as the difference between the recorded time of opening the note and the recorded time the note was signed in the EPIC electronic health record system.

SECONDARY OUTCOMES:
Number of notes completed after shift | within 1 week of posting note
  Shifts are 7 a.m. - 7 p.m for doctors assigned to daytime work. We defined a note completed after shift as any note with a signed time that is after 7 p.m. on the day of a shift worked.
Physician Satisfaction with EPIC Electronic Health Record | at baseline, 15-20 shifts, and 35-40 shifts
  We asked the participants this question:
  How comfortable are you specifically using the EPIC program for inpatient practice?" at baseline, midpoint (after working 15-20 shifts), and end of the study (after working 35-40 shifts).

CONTACTS AND LOCATIONS:
Overall Officials: Leena Jalota, MBBS, Principal Investigator — Reading Health System; Anthony A Donato, MD MHPE, Study Director — Reading Health System
Locations (1):
- Reading Health System, West Reading, Pennsylvania, United States